CLINICAL TRIAL: NCT00128011
Title: A Safety and Immunogenicity Study of a New Formulation of the Locally-Produced Bivalent Killed, Whole-Cell Oral Cholera Vaccine in Vietnamese Subjects
Brief Title: Safety and Immunogenicity of a New Formulation of a Bivalent Killed, Whole-Cell Oral Cholera Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: National Institute of Hygiene and Epidemiology, Vietnam (Other); Göteborg University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: C-12
Record Dates: First submitted 2005-08-08; First posted 2005-08-09 (Estimated); Last update posted 2006-11-10 (Estimated); Status verified 2006-11

CONDITIONS: Cholera
Keywords: watery diarrhea; cholera vaccine
MeSH Terms: conditions — Cholera

INTERVENTIONS:
Biological: killed oral cholera vaccine

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of a new formulation of a locally-produced bivalent, (O-1 and O-139) killed whole cell oral cholera vaccine among Vietnamese adults.

DETAILED DESCRIPTION:
Cholera remains to be a serious public health problem worldwide. In the mid-1980s following technology transfer from Sweden, Vietnamese scientists developed and produced an oral killed monovalent cholera vaccine for Vietnam's public health programs. A 2-dose regimen of this vaccine has been shown to be safe and efficacious. Subsequently, a bivalent vaccine was developed containing the newly emergent O139 V. cholerae. This vaccine has several advantages over the existing Swedish vaccine. It confers protection against the El Tor biotype in younger children, is considerably less expensive, does not require a buffer during administration and does not require strict cold chain requirements. However, this vaccine is not licensed for use in countries other than Vietnam. In order to make this vaccine available to other countries, the IVI has provided technical assistance to produce this vaccine following the WHO Good Manufacturing Practices standards. A new formulation of the current oral cholera vaccine was produced following these guidelines. Since this vaccine is slightly different from the previous vaccine, a study is necessary to demonstrate safety and immunogenicity for local licensure and larger Phase III studies in other countries.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-pregnant adults
* Available in the study area for 1 month

Exclusion Criteria:

* Diarrhea for the past week
* Antibiotic use in the past week
* Intake of anti-diarrheal medicines in the past week
* One or more episodes of diarrhea or abdominal pain lasting for 2 weeks during the past 6 months
* Abdominal pain, nausea, vomiting, loss of appetite or generalized ill feeling for the past 24 hours
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150
Dates: Start 2005-05; Study Completion 2005-06

PRIMARY OUTCOMES:
Adverse events
Serum Vibriocidal antibody response

CONTACTS AND LOCATIONS:
Overall Officials: Dang Duc Anh, PhD, Principal Investigator — National Institute of Hygiene and Epidemiology, Vietnam
Locations (1):
- National Institute of Hygiene and Epidemiology, Hanoi, Vietnam

REFERENCES:
- [Result] Anh DD, Canh DG, Lopez AL, Thiem VD, Long PT, Son NH, Deen J, von Seidlein L, Carbis R, Han SH, Shin SH, Attridge S, Holmgren J, Clemens J. Safety and immunogenicity of a reformulated Vietnamese bivalent killed, whole-cell, oral cholera vaccine in adults. Vaccine. 2007 Jan 22;25(6):1149-55. doi: 10.1016/j.vaccine.2006.09.049. Epub 2006 Sep 29. PMID 17055622